CLINICAL TRIAL: NCT00600561
Title: Biobehavioral Effects of Mindfulness-Based Stress Reduction in HIV
Brief Title: Mindfulness Meditation Training in HIV
Acronym: MBSR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Hector F. Myers, PhD, UCLA Department of Psychology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBSR-HIV-Trial-Seedgrant; M01RR000865 (NIH)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: HIV Infections
Keywords: meditation; mindfulness; HIV; CD4; Complementary Therapies
MeSH Terms: conditions — HIV Infections | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Day MBSR (Active Comparator): One-day condensed MBSR class
  Interventions: Behavioral: MBSR
- 8-week MBSR (Experimental): 8-week Mindfulness-Based Stress Reduction Intervention
  Interventions: Behavioral: MBSR

INTERVENTIONS:
Behavioral: MBSR — Mindfulness-Based Stress Reduction Intervention
  Other Names: mindfulness meditation; attention training

SUMMARY:
The purpose of this study is to investigate whether Mindfulness-Based Stress Reduction (MBSR) vs a one-day MBSR seminar improves immune (CD4+ T lymphocytes) and virological (HIV viral load) status in HIV-1 infected adults. The secondary goal of the study is to determine if MBSR vs a one-day MBSR seminar improves self-reported HIV-related quality of life.

DETAILED DESCRIPTION:
Mindfulness meditation, which is described as a process of bringing awareness to moment-to-moment experience, has been receiving substantial scientific attention as a process that can be stress and health protective (Brown, Ryan, & Creswell, 2007). Recent reviews by Baer (2003), Bishop (2002), and Grossman et al (2004) support the effectiveness of the standardized and manualized MBSR program in reducing stress and functional disability in a variety of chronic illnesses, although no studies have tested if MBSR impacts clinical markers of HIV, although some evidence suggests that MBSR improves some markers of innate immunity and quality of life in HIV-infected adults (see Robinson, Mathews, & Witek-Janusek, 2003). In this study, we propose to extend this work by investigating the impact of this intervention on biological and functional health status in HIV-positive adults.

We propose to determine whether the 8-week MBSR program is more effective than a one-day MBSR seminar in: (1) maintaining immune resistance in HIV infection (i.e. maintaining counts of CD4+ T lymphocytes and reducing HIV viral load), and (2) improving HIV-related quality of life. Additional analyses will test for a dose-response effect of MBSR by examining if MBSR class attendance and daily meditation practice are associated with the primary and secondary outcomes. These aims will be tested in a sample of 50 HIV-positive adults that is diverse with respect to ethnicity, gender and sexual orientation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed HIV for > 6 months
* English speaking
* 18 years old or older
* Indicate some distress (>4 on the Patient Health Questionnaire-9)
* Willing to be randomized

Exclusion Criteria:

* Any substance abuse or treatment for a psychiatric disorder in the past 30 days
* Currently diagnosed with AIDS or had CD4+ T lymphocytes <200 cells
* Hepatitis (A, B, or C)
* Indicate a regular mind-body practice (e.g., yoga, meditation) in the past six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
CD4+ T lymphocytes (counts) | Pre-test and post-test

SECONDARY OUTCOMES:
HIV-related Quality of Life | Pre-test and post-test
HIV viral load | Pre-test and post-test

CONTACTS AND LOCATIONS:
Overall Officials: Hector F Myers, PhD, Principal Investigator — University of California, Los Angeles; J. David Creswell, PhD, Study Director — Cousins Center for Psychoneuroimmunology, UCLA
Locations (1):
- Cousins Center for Psychoneuroimmunology, UCLA, Los Angeles, California, United States

REFERENCES:
- [Background] Hinkin CH, Barclay TR, Castellon SA, Levine AJ, Durvasula RS, Marion SD, Myers HF, Longshore D. Drug use and medication adherence among HIV-1 infected individuals. AIDS Behav. 2007 Mar;11(2):185-94. doi: 10.1007/s10461-006-9152-0. PMID 16897351
- [Background] Creswell JD, Way BM, Eisenberger NI, Lieberman MD. Neural correlates of dispositional mindfulness during affect labeling. Psychosom Med. 2007 Jul-Aug;69(6):560-5. doi: 10.1097/PSY.0b013e3180f6171f. Epub 2007 Jul 18. PMID 17634566
- [Derived] Creswell JD, Myers HF, Cole SW, Irwin MR. Mindfulness meditation training effects on CD4+ T lymphocytes in HIV-1 infected adults: a small randomized controlled trial. Brain Behav Immun. 2009 Feb;23(2):184-8. doi: 10.1016/j.bbi.2008.07.004. Epub 2008 Jul 19. PMID 18678242